CLINICAL TRIAL: NCT05130086
Title: A Phase 2 Open-Label Study to Evaluate the Safety and Pharmacokinetics of Oral Islatravir Once-Monthly in Trans and Gender Diverse Individuals on Gender-Affirming Hormone Therapy and at Low-Risk for HIV-1 Infection
Brief Title: A Study of Islatravir (MK-8591) in Trans and Gender Diverse Participants (MK-8591-035)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Business Reasons
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 8591-035; MK-8591-035 (Other: Merck)
Record Dates: First submitted 2021-11-10; First posted 2021-11-22 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Human Immunodeficiency Virus (HIV) Infections
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Infections | interventions — islatravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Islatravir (Experimental): 60 mg Islatravir taken orally in tablet form once monthly for up to 24 weeks
  Interventions: Drug: Islatravir

INTERVENTIONS:
Drug: Islatravir — 60 mg Islatravir taken orally in tablet form once monthly for up to 24 weeks
  Other Names: MK-8591

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of Islatravir (ISL) in trans and gender diverse (TGD) participants who are receiving gender-affirming hormone therapy (GAHT) and are at low-risk for human immunodeficiency virus 1 (HIV-1) infection.

ELIGIBILITY:
Inclusion Criteria:

* Is confirmed HIV-uninfected based on negative HIV-1/HIV-2 test result before allocation to study intervention.
* Is on stable GAHT and does not intend to change therapy through Week 4 of the study.
* Has a low-risk of HIV infection.
* Identifies with a gender that is different from that assigned at birth.
* A participant assigned female at birth is eligible if not pregnant or chest-feeding and is not of childbearing potential (POCBP) or: Is a POCBP and using an acceptable contraceptive method, or be abstinent from penile-vaginal intercourse with an individual capable of producing sperm (abstinent on a long term and persistent basis); a POCBP must have a negative highly sensitive pregnancy test ([urine or serum] as required by local regulations) within 24 hours before the first dose of study intervention; If a urine test cannot be confirmed as negative (e.g, an ambiguous result), a serum pregnancy test is required. In such cases, the participant must be excluded from participation if the serum pregnancy result is positive; the investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a participant assigned female at birth with an early undetected pregnancy; contraceptive use by participant assigned female at birth should be consistent with local regulations.

Exclusion Criteria:

* Has known current or chronic history of liver disease (e.g, non-alcoholic or alcoholic steatohepatitis) or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome, asymptomatic gallstones, or cholecystectomy), unless the participant has stable liver function tests and no evidence of hepatic synthetic dysfunction.
* Has a history of malignancy within 5 years of screening except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or in situ anal cancers.
* Has taken cabotegravir, lenacapavir, or any other long-acting HIV prevention product at any time (past or current use).
* Is currently participating in or has participated in a clinical study with an investigational compound or device, within 30 days before Day 1 through the duration of the study.
* Is expecting to conceive or donate eggs at any time during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants will include anyone who identifies with a gender that is different from the sex assigned at birth (e.g., transgender woman, transgender man, gender nonbinary, etc.), including those with differences in sex development (sometimes called intersex).
Enrollment: 0 (Actual)
Dates: Start 2022-10-17 (Estimated); Primary Completion 2024-03-25 (Estimated); Study Completion 2024-03-25 (Estimated)

PRIMARY OUTCOMES:
Participants with one or more adverse events (AEs) | Up to 26 weeks
  Number of participants with one or more AEs will be reported.
Participants with an AE leading to discontinuation of study intervention | Up to 20 weeks
  Number of participants with an AE leading to discontinuation of study intervention will be reported.

SECONDARY OUTCOMES:
Area Under the Curve (AUC) of plasma islatravir (ISL) | Pre-dose on Day 1; any time on Weeks 1, 2 and 3; pre-dose on Weeks 4, 8, 12, 16, 20; any time on Week 24
  Area Under the Curve from time 0 to 672 hours post-dose (AUC0-672hr) of plasma islatravir (ISL) will be reported.
Maximum concentration (Cmax) of plasma ISL | Pre-dose on Day 1; any time on Weeks 1, 2 and 3; pre-dose on Weeks 4, 8, 12, 16, 20; any time on Week 24
  Maximum concentration (Cmax) of plasma ISL will be reported.
Trough concentration (Ctrough) of plasma ISL | Pre-dose on Day 1; any time on Weeks 1, 2 and 3; pre-dose on Weeks 4, 8, 12, 16, 20; any time on Week 24
  Trough concentration (Ctrough) of plasma ISL will be reported.
Apparent terminal half-life (t1/2) of plasma ISL | Pre-dose on Day 1; any time on Weeks 1, 2 and 3; pre-dose on Weeks 4, 8, 12, 16, 20; any time on Week 24
  Apparent terminal half-life (t1/2) of plasma ISL will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php